CLINICAL TRIAL: NCT02574754
Title: Assessment of 2012 Bioequivalence Standards for Narrow Therapeutic Index Drugs: a Study With Warfarin
Brief Title: Assessment of 2012 Bioequivalence Standards for Warfarin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 15-17226
Record Dates: First submitted 2015-09-09; First posted 2015-10-14 (Estimated); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Healthy
Keywords: warfarin; pharmacokinetics; bioequivalence; healthy volunteer
MeSH Terms: interventions — Warfarin; Vitamin B 6

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- warfarin (Experimental): Subjects will receive a single dose of warfarin 10 mg PO at each of 3 visits. The study days will be separated by at least 14 days to allow adequate time for the drug to reach washout.
  Interventions: Drug: warfarin

INTERVENTIONS:
Drug: warfarin — warfarin 10 mg PO x 1
  Other Names: Coumadin; Jantoven

SUMMARY:
The purpose of this study is to assess the 2012 bioequivalence statistical criteria for warfarin, a narrow therapeutic index drug, set forth in the draft guidance issued by the Food and Drug Administration (FDA).

DETAILED DESCRIPTION:
This study is a reasonable starting point to assess the appropriateness of the 2012 FDA bioequivalence (BE) statistical criteria for narrow therapeutic index drugs (NTIDs). The idea stems from an earlier study conducted in Dr. Benet's lab with the drug furosemide. The furosemide study yielded triplicate data that were unable to purely meet the BE statistical criteria set forth by the FDA due to the inherent study design. Furosemide is not an NTID to be considered by the FDA for BE studies, however. Hence, the investigators have proposed a new study to assess the BE statistical criteria with warfarin, an NTID with a draft guidance issued by the FDA. By providing the reference product (brand name warfarin) three times to each study participant and recording the relevant pharmacokinetic parameters for BE (AUC and Cmax), the investigators can make three comparisons between the data (R1 and R2 vs. R2 and R3; R1 and R2 vs. R1 and R¬3; R2 and R3 vs. R1 and R3).

The investigators have three concerns that can be tested here.

1. Will normal within subject variability potentially lead to inequivalence of the reference product using the new NTID BE regulations?
2. Is it possible that the BE interval could be less than the United States Pharmacopeia (USP) content uniformity limits for warfarin?
3. Provide a comparison of the within-subject variance for the 2.5 ratio comparison.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18-60 years
* Healthy adult without active medical problems or chronic diseases based on medical history, physical exam, and laboratory results
* BMI 18.5-32 kg/m2
* Ceased all medications 2 weeks prior to start of study and during study enrollment (includes drugs of abuse, prescription medications, and over-the-counter (OTC) medications [exception: acetaminophen])
* Maintain adequate birth control independent of hormonal contraceptive use throughout study
* Provide written informed consent to take part in and comply with the requirements of the study
* Speak, read, and understand English
* Avoid alcohol, caffeine, and orange juice from 6pm the night before the study day until the completion of the study day
* Avoid contact sports and/or other activities with significant risk of trauma injury for 7 days after each study day
* Do not eat food or consume beverages at least 8 hours before medication dosing
* Present with wild type VKORC1, VKORC-1639G>A and wild type CYP2C9 genotype

Exclusion Criteria:

* Subjects on prescription or chronic OTC medications (including hormonal contraceptives)
* Subjects with known allergy to warfarin
* Subjects with a history of or diagnosis of hemorrhagic tendencies or blood dyscrasias
* Subjects with liver failure or liver function tests (LFTs) > 2x upper limit normal
* Subjects with clinically significant elevations of international normalized ratio (INR), prothrombin time (PT), partial thromboplastin time (PTT), serum creatinine (Scr), blood urea nitrogen (BUN), or other screening laboratory tests as determined by study physician
* Subjects with hematocrit (Hct) < 30 mg/dL
* Subjects with history of GI bleed or peptic ulcer disease
* Subjects with recent history of trauma
* Subjects with recent history of or upcoming plan for surgery
* Subjects who smoke tobacco
* Subjects with ongoing alcohol use
* Subjects with ongoing illegal drug use
* Subjects who are pregnant, attempting to become pregnant, or lactating
* Subjects who are unable to maintain adequate birth control during the study
* Subjects who are unable to follow protocol instructions or criteria
* Subjects with genotypes that are not wild type VKORC1, VKORC-1639G>A and wild type CYP2C9

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2016-05; Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
S- and R- enantiomers of warfarin (S-warfarin, R-warfarin) Area Under the Plasma Concentration-Time Curve (AUC) from 0 to 72 hours | 0 to 72 hours after warfarin dosing
  The primary outcome measure will be warfarin area-under-the-concentration-time curve (AUC) values from zero to seventy-two (0-72) hours. Values from the Experimental Arm (warfarin) of each the 3 study periods will be compared against each other and analyzed for intra-individual variability and tested for bioequivalence using the new narrow therapeutic index drug (NTID) regulations. Blood collection at 0, 1, 2, 3, 4, 6, 8, 12 hours after warfarin dosing.

SECONDARY OUTCOMES:
S- and R- enantiomers of warfarin (S-warfarin, R-warfarin) Area Under the Plasma Concentration-time Curve (AUC) from time zero to infinity hours | 0 to 8 weeks after warfarin dosing
  A secondary outcome measure will be warfarin area-under-the-concentration-time curve (AUC) values from zero to infinite time (0-inf) where infinite time represents the duration of the study (8 weeks). Values from the Experimental Arm (warfarin) of each the 3 study periods will be compared against each other and analyzed for intra-individual variability and tested for bioequivalence using the new narrow therapeutic index drug (NTID) regulations. Analysis of all concentration-time data; blood collection at 0, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours after warfarin dosing.
Maximum Plasma Concentration (Cmax) of S-warfarin and R-warfarin | 0 to 72 hours after warfarin dosing
  A secondary outcome measure will be maximum plasma concentration (Cmax). Values from the Experimental Arm (warfarin) of each the 3 study periods will be compared against each other and analyzed for intra-individual variability and tested for bioequivalence using the new narrow therapeutic index drug (NTID) regulations. Blood collection 0, 1, 2, 4, 6, 8, 12, 24, 48, and 72 hours after warfarin dosing.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Z Benet, PhD, Principal Investigator — University of California, San Francisco; Lynda A Frassetto, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States